CLINICAL TRIAL: NCT05608525
Title: Effects of Transcranial Direct Current Stimulation on Upper Limb Motor Rehabilitation in Chronic Stroke Patients
Brief Title: Upper Limb tDCS in Chronic Stroke Patients (NOURISH)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2022/00686
Record Dates: First submitted 2022-11-01; First posted 2022-11-08 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: Stroke
Keywords: stroke; motor recovery; transcranial direct current stimulation; corticospinal excitability; neuromodulation
MeSH Terms: conditions — Stroke | interventions — Transcranial Direct Current Stimulation; Hand Strength

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to receive one of the followings:
  * Group 1 will receive 1 mA anodal tDCS stimulation to the ipsilesional M1 of cortical representation of the affected upper limb;
  * Group 2 to receive 1mA anodal tDCS to the contralesional premotor cortex;
  * Group 3 to receive sham tDCS stimulation with anode placed over the scalp area corresponding to ipsilesional M1.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participant and outcome assessor will be blinded to the tDCS stimulation protocol that they will be receiving.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Anodal tDCS stimulation to the ipsilesional M1 (Experimental): Participant will receive 1 mA anodal tDCS stimulation to the ipsilesional M1 of cortical representation of the affected upper limb.
  Cathode will be used as reference electrode and placed over the supraorbital area contralateral to the anode. tDCS stimulation will be conducted daily for 20 sessions in consecutive days in the 4th month after stroke, with each session lasting for 20 minutes and combined with online occupational therapy training.
  Interventions: Device: transcranial current stimulation; Behavioral: GRASP
- Anodal tDCS to the contralesional premotor cortex (Experimental): Participant will receive 1mA anodal tDCS to the contralesional premotor cortex. Cathode will be used as reference electrode and placed over the supraorbital area contralateral to the anode. tDCS stimulation will be conducted daily for 20 sessions in consecutive days in the 4th month after stroke, with each session lasting for 20 minutes and combined with online occupational therapy training.
  Interventions: Device: transcranial current stimulation; Behavioral: GRASP
- Sham tDCS (Sham Comparator): Participant will receive sham tDCS stimulation with anode placed over the scalp area corresponding to ipsilesional M1.
  Cathode will be used as reference electrode and placed over the supraorbital area contralateral to the anode. tDCS stimulation will be conducted daily for 20 sessions in consecutive days in the 4th month after stroke, with each session lasting for 20 minutes and combined with online occupational therapy training.
  Interventions: Device: transcranial current stimulation; Behavioral: GRASP

INTERVENTIONS:
Device: transcranial current stimulation — A trained research staff or physician will perform tDCS to the subject. Direct current will be delivered by a battery-operated, constant current stimulator, through 2 rubber electrodes embedded in a pair of saline-soaked sponge bag. Stimulation intensity will be ramped up to 1 mA over 30 seconds and maintain at 1 mA for 20 minutes, and then ramped down to 0 mA over 30 seconds.
Behavioral: GRASP — A standardized occupational therapy- GRASP will be performed daily together with tDCS over the period between the Pre Assessment and the Post Assessment. GRASP exercise will be administered concurrently with or immediately after tDCS stimulation. GRASP is a self-directed arm and hand exercise program for which is supervised by a therapist, but done independently by the participant (and with their family if possible). GRASP has been shown to improve arm and hand function and strength in stroke patients in community [22-27]. The versions of the program- Home GRASP will be used. All occupational tasks will be selected from the GRASP task pool and be progressed according to the GRASP protocol (https://neurorehab.med.ubc.ca/grasp). Each GRASP session will take about 1 hour. A total of 20 GRASP sessions will be administered.

SUMMARY:
This study is a randomized double-blinded trial investigating the effect of Transcranial Direct Current stimulation (tDCS) on upper limb motor function rehabilitation in chronic stroke patients.

51 subjects will be recruited from National University Hospital (NUH) and be randomized to receive one of the followings:

* Group 1 will receive 1 mA anodal tDCS stimulation to the ipsilesional M1 of cortical representation of the affected upper limb;
* Group 2 to receive 1mA anodal tDCS to the contralesional premotor cortex;
* Group 3 to receive sham tDCS stimulation with anode placed over the scalp area corresponding to ipsilesional M1.

tDCS will be performed once a day together with standardized occupational therapy (GRASP) for 20 sessions within 30 days. Group 1 and Group 2 will receive tDCS for 20 minutes during each session, while Group 3 only receives the current stimulation for 20 seconds. GRASP will be performed daily together with tDCS, either concurrently with or immediately after tDCS stimulation.

The outcome measures will be measured at baseline, after intervention and 1 month after intervention, including:

1. TMS measurement of corticospinal excitability;
2. functional MRI scan;
3. High density EEG (HD-EEG) evaluation;
4. Clinical measures on upper limb motor function;
5. Cognitive tests.

DETAILED DESCRIPTION:
This study is a randomized double-blinded trial investigating the effect of Transcranial Direct Current stimulation (tDCS) on upper limb motor function rehabilitation in chronic stroke patients.

51 subjects will be recruited from National University Hospital (NUH). Once subject is identified to be eligible for the study and is agreeable to participate into the study, the following will be measured/performed:

1. TMS measurement of corticospinal excitability: resting motor threshold and/or active motor threshold, intracortical facilitation, short interval intracortical inhibition, silent period.
2. MRI scan: Participants will go through the following image acquisition procedures at NUS TMR (Centre for Translational MR Research): 1) a functional MRI scans for brain activity together with motor task. 2) a 3D MPRAGE sequence for brain structure. 3) an advanced multishell high-resolution diffusion MRI for characterizing brain microstructure and extracellular space. 4) a FLAIR scan to measure white matter hyperintensity. Both functional and anatomical image acquisition will be undertaken using but not limited to gradient echo EPI sequence or its modified version (Feinberg & Setsompop, 2013). Signal stability during imaging is assured by a daily prescan QC routine. Contrast MRI will not be performed in this study. The MRI scan will take about 1 hours. The whole procedure including briefing and preparation will be about 1.5 hours.
3. High density EEG (HD-EEG) evaluation of the electrical activity of the brain.
4. Clinical measures on upper limb motor function:

   * upper extremity portion of Fugl-Meyer Assessment (UE-FMA)
   * Action Research Arm test (ARAT)
   * Modified Ashworth scale for spasticity (MAS)
   * Isometric elbow flexion strength
   * Handgrip strength
5. Cognitive tests:

   * Digit Span Task
   * Digit Symbol Modalities Task
   * Trail-making test (TMT)-A &B
   * Clock-Drawing Test (CDT)
   * Controlled Oral Word Association Test (COWAT) -animals & FAS
   * Mini-Mental State Exam (MMSE)
   * Rey Auditory Verbal Learning Test (RAVL)
   * Spatial span forward/backward test
   * Visuospatial Paired Associate Learning (VPA)
6. Randomization: Subject will be randomized into 3 groups using Microsoft Excel, to receive different types of stimulation:

   * Group 1 will receive 1 mA anodal tDCS stimulation to the ipsilesional M1 of cortical representation of the affected upper limb;
   * Group 2 to receive 1mA anodal tDCS to the contralesional premotor cortex;
   * Group 3 to receive sham tDCS stimulation with anode placed over the scalp area corresponding to ipsilesional M1.

The assessor of the outcome measures and subject will be blinded to the tDCS intervention that subject will be receiving.

After the outcome measures (Pre Assessment) are done, tDCS will be performed once a day together with standardized occupational therapy (GRASP) for 20 sessions within 30 days.

Direct current will be delivered by a battery-operated, constant current stimulator (HDCstim, Magstim), through 2 rubber electrodes embedded in a pair of saline-soaked sponge bag. Stimulation intensity will be ramped up to 1 mA over 30 seconds and maintain at 1 mA for 30 minutes, and then ramped down to 0 mA over 20 seconds. Sham-tDCS was delivered by similarly ramping up to 1 mA but maintained for only 20 seconds to give subjects the same scalp sensation, before ramping down. Cathode for all 3 tDCS groups will be used as reference electrode and placed over the supraorbital area contralateral to the anode.

Three options will be provided for subject to decide where the 20 sessions of tDCS intervention will be performed. Subject could choose either 1 option or "mixed option".

1. At NUH: which is recommended by the study team.
2. At home and assisted by caregiver: For subject's convenience and to minimize the number of hospital visits especially during unforeseen circumstance like COVID outbreak, subject is allowed to bring tDCS device (Stimulator only) back to use at home after the caregiver is properly trained. Literature has shown that administration of tDCS at home by patient and caregiver is feasible and safe [13].

   The protocol details of tDCS home usage is elaborated in the document "Study Protocol".
3. At home and assisted by research staff: Research staff can go subject's home to perform tDCS stimulation. In this case, tDCS stimulator will be kept by research staff.

A standardized occupational therapy- GRASP will be performed daily together with tDCS over the period between the Pre Assessment and the Post Assessment. GRASP exercise will be administered concurrently with or immediately after tDCS stimulation. GRASP is a self-directed arm and hand exercise program for which is supervised by a therapist, but done independently by the participant (and with their family if possible). GRASP has been shown to improve arm and hand function and strength in stroke patients in community [22-27]. The versions of the program- Home GRASP will be used. All occupational tasks will be selected from the GRASP task pool and be progressed according to the GRASP protocol (https://neurorehab.med.ubc.ca/grasp). Each GRASP session will take about 1 hour. A total of 20 GRASP sessions will be administered.

The same outcome measures will be performed again after 20 sessions of tDCS (Post Assessment), and 1 month after the tDCS intervention (Follow-up Assessment), except that MRI scan will not be performed at Post Assessment.

ELIGIBILITY:
Inclusion Criteria:

* Age 21-80 years old;
* First ever stroke, 6 months to 2 years after stroke onset;
* ARAT≤42

Exclusion Criteria:

1. Pregnancy;
2. Any metal implants inside the body that are contraindications of MRI scan;
3. cardiac pacemakers;
4. History of epilepsy;
5. Sensorimotor disturbance due to other causes other than stroke;
6. Claustrophobia;
7. Uncontrolled medical conditions including hypertension, diabetes mellitus and unstable angina;
8. Major depression and a history of psychotic disorders;
9. Terminal diagnosis with life expectancy <=1 year. Any metal implants inside the body that are contraindications of MRI scan;

3. cardiac pacemakers; 4. History of epilepsy; 5. Sensorimotor disturbance due to other causes other than stroke; 6. Claustrophobia; 7. Uncontrolled medical conditions including hypertension, diabetes mellitus and unstable angina; 8. Major depression and a history of psychotic disorders; 9. Terminal diagnosis with life expectancy <=1 year.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Estimated)
Dates: Start 2023-02-16 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Cortical excitability measured by Transcranial Magnetic Stimulation (TMS) | Month 0
  measures of cortical excitability for those without TMS contraindications
Cortical excitability measured by Transcranial Magnetic Stimulation (TMS) | Month 1
  measures of cortical excitability for those without TMS contraindications
Cortical excitability measured by Transcranial Magnetic Stimulation (TMS) | Month 2
  measures of cortical excitability for those without TMS contraindications
neural excitability measured by Magnetic resonance imaging (MRI) scan | Month 0
  Participants will go through one of the following image acquisition procedures 1) a functional MRI scans for brain activity together with motor task. 2) a 3D MPRAGE sequence for brain structure. 3) an advanced multishell high-resolution diffusion MRI for characterizing brain microstructure and extracellular space. 4) a FLAIR scan to measure white matter hyperintensity. Both functional and anatomical image acquisition will be undertaken using but not limited to gradient echo EPI sequence or its modified version.
neural excitability measured by Magnetic resonance imaging (MRI) scan | Month 2
  Participants will go through one of the following image acquisition procedures 1) a functional MRI scans for brain activity together with motor task. 2) a 3D MPRAGE sequence for brain structure. 3) an advanced multishell high-resolution diffusion MRI for characterizing brain microstructure and extracellular space. 4) a FLAIR scan to measure white matter hyperintensity. Both functional and anatomical image acquisition will be undertaken using but not limited to gradient echo EPI sequence or its modified version.
neural excitability measured by electroencephalogram (EEG) | Month 0
  High density EEG (electroencephalogram) evaluation of the electrical activity of the brain
neural excitability measured by electroencephalogram (EEG) | Month 1
  High density EEG (electroencephalogram) evaluation of the electrical activity of the brain
neural excitability measured by electroencephalogram (EEG) | Month 2
  High density EEG (electroencephalogram) evaluation of the electrical activity of the brain
upper extremity motor function using Fugl-Meyer scale | Month 0
  Upper limb function, Minimum score 0, Maximum score 66, the higher the score the better the upper limb function.
upper extremity motor function using Fugl-Meyer scale | Month 1
  Upper limb function, Minimum score 0, Maximum score 66, the higher the score the better the upper limb function.
upper extremity motor function using Fugl-Meyer scale | Month 2
  Upper limb function, Minimum score 0, Maximum score 66, the higher the score the better the upper limb function.
Action Research Arm Test | Month 0
  Test for upper extremity performance (coordination, dexterity and functioning). Minimum score 0, Maximum score 57, the higher the score the better the upper limb function.
Action Research Arm Test | Month 1
  Test for upper extremity performance (coordination, dexterity and functioning). Minimum score 0, Maximum score 57, the higher the score the better the upper limb function.
Action Research Arm Test | Month 2
  Test for upper extremity performance (coordination, dexterity and functioning). Minimum score 0, Maximum score 57, the higher the score the better the upper limb function.
Modified Ashworth scale for spasticity (MAS) | Month 0
  Test for muscle spasticity. 6 point scale, Scores range from 0 to 4 (namely 0, 1, 1+, 2, 3 and 4), where lower scores represent normal muscle tone and higher scores represent spasticity or increased resistance to passive movement.
Modified Ashworth scale for spasticity (MAS) | Month 1
  Test for muscle spasticity. 6 point scale, Scores range from 0 to 4 (namely 0, 1, 1+, 2, 3 and 4), where lower scores represent normal muscle tone and higher scores represent spasticity or increased resistance to passive movement.
Modified Ashworth scale for spasticity (MAS) | Month 2
  Test for muscle spasticity. 6 point scale, Scores range from 0 to 4 (namely 0, 1, 1+, 2, 3 and 4), where lower scores represent normal muscle tone and higher scores represent spasticity or increased resistance to passive movement.

CONTACTS AND LOCATIONS:
Overall Officials: Effie Chew, MBBS, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore